CLINICAL TRIAL: NCT00803751
Title: A Comparison of the Infant Truview EVO2 Video Laryngoscope and the Macintosh Laryngoscope in Pediatric Patients
Acronym: Truview
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Maria Matuszczak, Professor - Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Infant Truview
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2011-03

CONDITIONS: Laryngoscopy
Keywords: Laryngoscopy [E04.580.373]

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Truview intubation (Experimental): Receive laryngoscopy with Truview first and is immediately followed by laryngoscopy and intubation with Macintosh
  Interventions: Device: Truview EVO2 laryngoscope
- Macintosh intubation (Active Comparator): Macintosh blade will be used first followed by laryngoscopy and intubation with the truview
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: Truview EVO2 laryngoscope — will use the Truview laryngoscope instead of the traditional Macintosh laryngoscope
  Arms: Truview intubation
Device: Macintosh laryngoscope — Intubation using the traditional Macintosh laryngoscope
  Arms: Macintosh intubation

SUMMARY:
This study is intended to examine the effectiveness of a new type of laryngoscope, the Truview EVO2, in an infant patient population. They device will be tested against the current clinical standard, the Macintosh laryngoscope, in patients undergoing surgery at our hospital in terms of ease of use, view obtained of the vocal cords, and ability to place an endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than one year
2. Requiring general anesthesia and orotracheal intubation
3. Weight less than 10 kg
4. ASA class 1-3

Exclusion Criteria:

1. Documented difficult airway
2. Facial deformities

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Matuszczak, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital - Texas Medical Center, Houston, Texas, United States

REFERENCES:
- See also: Truphatek - Manufacturer's website — http://www.truphatek.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from pediatric day surgery.
Pre-assignment Details: There were 11 patients excluded from the trial due to incomplete data.
Groups:
- Truview Intubation First Then With Macintosh: Receive laryngoscopy with Truview blade first and is immediately followed by laryngoscopy and intubation with Macintosh blade
- Macintosh Intubation First Followed by Truview Intubation: Use the Macintosh laryngoscope first immediately followed by laryngoscopy and intubation with the Truview laryngoscope
Period: Overall Study
Arm/Group | Truview Intubation First Then With Macintosh | Macintosh Intubation First Followed by Truview Intubation
Started | 26 | 23
Completed | 26 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Truview Intubation First Then With Macintosh | Macintosh Intubation First Followed by Truview Intubation | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 23 | 49
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 6.35 (3.1) | 6.42 (3.2) | 6.39 (3.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 26 | 23 | 49

OUTCOME MEASURES:

1. Primary Outcome: Quality of Laryngeal View Obtained on Comarck Lehane Classification
Description: The view obtained when we do laryngoscopy. The Comarck Lehane classification is as follows: 1) Most of the glottis is seen; 2a) Only the posterior part of the glottis is visible; 2b) The epiglottis is visible, but none of the glottis can be seen; 3) Not even the epiglottis is visible.
Time Frame: during laryngoscopy prior to intubation. Few minutes before intubation
Measure: Number; unit: Participants
Groups:
- Truview: This group has data for all the truview intubations
- Mac Blade: This groups has data with all the mac blade intubations
Arm/Group | Truview | Mac Blade
Number analyzed (Participants) | 26 | 23
Participants
  1 | 21 | 13
  2a | 3 | 5
  2b | 1 | 4
Statistical Analysis 1: Comparison: Truview vs Mac Blade; Test type: Superiority or Other; p = 0.17, Fisher Exact

2. Primary Outcome: Number of Intubation Attempts
Description: Number of participants with the indicated number of intubation attempts (1/2/3)
Time Frame: during intubation prior to surgery
Measure: Number; unit: Participants
Arm/Group | Truview | Mac Blade
Number analyzed (Participants) | 26 | 23
Participants
  1 | 17 | 23
  2 | 4 | 2
  3 | 2 | 1
Statistical Analysis 1: Comparison: Truview vs Mac Blade; Test type: Superiority or Other; p = 0.45, Fisher Exact

3. Secondary Outcome: Time Taken for Intubation
Time Frame: throughout the intubation procedure
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Truview | Mac Blade
Number analyzed (Participants) | 26 | 23
seconds | 25.23 (11.09) | 28.33 (12.67)
Statistical Analysis 1: Comparison: Truview vs Mac Blade; Test type: Superiority or Other; p = 0.36, t-test, 2 sided

4. Secondary Outcome: POGO Score With 1st Laryngoscopy
Description: POGO score is the percent of glottic opening observed during laryngoscopy. 100% POGO score indicates a full view of glottic opening and 0% POGO score indicates no glottic opening.
Time Frame: Before patient is intubated (few minutes before intubation)
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Truview | Mac Blade
Number analyzed (Participants) | 26 | 23
Score | 93.65 (15.72) | 73.81 (23.34)
Statistical Analysis 1: Comparison: Truview vs Mac Blade; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

5. Primary Outcome: Quality of Laryngeal View Obtained With 2nd Laryngoscopy
Description: as for outcome 1
Time Frame: during laryngoscopy prior to intubation (few minutes prior to intubation)
Measure: Number; unit: Participants
Arm/Group | Truview | Mac Blade
Number analyzed (Participants) | 26 | 23
Participants
  1 | 10 | 21
  2a | 7 | 2
  2b | 9 | 0
Statistical Analysis 1: Comparison: Truview vs Mac Blade; Test type: Superiority or Other; p < 0.001, Fisher Exact

6. Secondary Outcome: POGO Score With 2nd Laryngoscopy
Description: as for outcome 4
Time Frame: Before patient is intubated
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Truview | Mac Blade
Number analyzed (Participants) | 26 | 23
Score | 74.3 (25.1) | 98.0 (8.94)
Statistical Analysis 1: Comparison: Truview vs Mac Blade; Test type: Superiority or Other; p = 0.0004, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Truview Intubation First Then With Macintosh | Macintosh Intubation First Followed by Truview Intubation
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No